CLINICAL TRIAL: NCT05484479
Title: Baduanjin-exercise Efficacy on Chronic Periodontal Disease in Elderly
Brief Title: Effect of Baduanjin Exercise on Chronic Periodontal Disease in Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003757
Record Dates: First submitted 2022-07-30; First posted 2022-08-02 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Chronic Periodontal Disease
MeSH Terms: conditions — Chronic Periodontitis | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercised group (Experimental): For 6 months, MeTS elderly (25 elderly) with chronic periodontal disease will be trained using sixty-minute Baduanjin training/exercise (5 times weekly)
  Interventions: Behavioral: Baduanjin training/exercise
- control group (No Intervention): For 6 months, MeTS elderly (25 elderly) with chronic periodontal disease will receive no training

INTERVENTIONS:
Behavioral: Baduanjin training/exercise — For 6 months, MeTS elderly (25 elderly) with chronic periodontal disease will be trained using sixty-minute Baduanjin training/exercise (5 times weekly)
  Arms: Exercised group

SUMMARY:
The metabolic syndrome (MetS) is a spectrum of conditions that increase the risk of cardiovascular disease and diabetes mellitus. The components of MetS include dysglycemia, visceral obesity, atherogenic dyslipidemia (elevated triglycerides and low levels of high-density lipoprotein) and hypertension. An association of periodontal disease and MetS has been suggested. This association is believed to be the result of systemic oxidative stress and an exuberant inflammatory response.

Physical activity is associated as a potential tool for reduction of periodontal disease prevalence. The frequency of physical activity is directly related to a low occurrence of periodontitis.

DETAILED DESCRIPTION:
For 6 months, MeTS elderly (25 elderly) with chronic periodontal disease will be involved in sixty-minute Baduanjin physical training (5 session weekly). Also, for 6 months, another MeTS elderly (25 elderly) with chronic periodontal disease will serve as a control non-trained group.

ELIGIBILITY:
Inclusion Criteria:

* fifty elderly with metabolic syndrome and chronic periodontal disease will be included
* both sexes will be included

Exclusion Criteria:

* smokers
* elderly engaged in physical activity programs
* any cardiovascular/respiratory diseases that obstacle the conduction of Baduanjin
* elderly on drug therapies for chronic periodontal disease

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — self-representation of gender identity
Enrollment: 50 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Periodontal disease index | It will be assessed after 6-month intervention
  it will assess periodontal health status

SECONDARY OUTCOMES:
Simplified oral hygiene index | It will be assessed after 6-month intervention
  it will assess oral hygiene/cleanliness status
Interleukin 1 beta | It will be after 6-month intervention
  it will be assessed in saliva
interleukin 6 | It will be assessed after 6-month intervention
  it will be assessed in saliva
superoxide dismutase | It will be assessed after 6-month intervention
  it will be assessed in saliva
total antioxidant status | It will be assessed after 6-month intervention
  it will be assessed in saliva

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Dokki, Egypt